CLINICAL TRIAL: NCT03732742
Title: Comparison of Mid-term Results of Total Correction of Tetralogy of Fallot Between Preservation of Pulmonary Valve and Trans-annular Patching
Brief Title: Comparison of Mid-term Results of Total Correction of TOF Between Preservation of PV and Trans-annular Patch.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shareef aldesoky shareef, Professor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TOF repair
Record Dates: First submitted 2018-10-22; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Tetrology of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOF repair with preservation of PV (Experimental): Surgical intervention by repair of Tetralogy of Fallot with preservation of pulmonary valve, recently interested has shifted to preserving the integrity of the pulmonary valve.
  Interventions: Procedure: TOF repair with trans-annular patch VS preservation of PV
- TOF repair with trans-annular patch (Experimental): Surgical intervention by repair of Tetralogy of Fallot with trans-annular patch, right ventricular hypertrophy, right ventricular dilatation and pulmonary vavle regurgitation has been recognized as one of the most important risk factors for both right and left ventricular performance after the repair of Tetralogy of Fallot.
  Interventions: Procedure: TOF repair with trans-annular patch VS preservation of PV

INTERVENTIONS:
Procedure: TOF repair with trans-annular patch VS preservation of PV — One group study

SUMMARY:
To compare of mid-term results of total correction of tetralogy of fallot between preservation of pulmonary valve and trans-annular patching , thus avoiding PV regurgitation during TOF repair , this will determine the value of this procedure over trans-annular patching regarding to right ventricular performance.

DETAILED DESCRIPTION:
Surgical repair of congenital lesions associated with right ventricular outflow tract obstruction frequently requires the destruction of pulmonary valve (PV) competents including the pulmonary annulas. The resulatnt pulmonary insufficiency may lead to late functional deterioration of right ventricular performance. Acute right ventricular dysfunction has been associated with poor pulmonary runoff, tricuspid valve regurgitaion and pulmonary hypertension. Preservation of PV comptence may prevent both early and late right ventricular failure. Total repair of tetralogy of fallot is a corrective surgical procedure that involves closure of the ventricular septal defect (VSD) and relief of right ventricular outflow tract (RVOT) obstruction. The surgeon must decide whether the right ventricular outflow tract size will be sufficient to allow for the entire cardiac output to traverse it without causing extreme elevation in right ventricular pressure or will go for trans-annular patch. Recently interest has shifted to preserving the integrity of the pulmonary valve annulus thus avoiding pulmonary valve regurgitation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective total correction of tetralogy of Fallot.
2. Any age group.
3. Normal pulmonay branches

Exclusion Criteria:

1. Patients associated with other congenital anomalies.
2. Regarding PV morphology, patients with pulmonary atresia , absence of PV.
3. Patients with anomalous coronary artery anatomy obstructs access to the RV
4. Extra-cardiac illness that is expected to limit survival to less than 5 years.e.g active hepatitis or significant hepatic or renal disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Gender | One week for preoperative assessment.
  Parameters will be measured include gender preoperatively
Body weight | One week for preoperative assessment.
  Parameters will be measured include body weight in kilograms preoperatively
Height | One week for preoperative assessment.
  Parameters will be measured include height in meters preoperatively
Oxygen saturation , RV function | One week for preoperative assessment.
  Parameters will be measured include Oxygen saturation level % , RV function by measure RV fractional area changes (RVFAC) % preoperatively
include median RVOT gradient and degree of PV stenosis | One week for preoperative assessment.
  Parameters will be measured include median RVOT gradient in mmhg , degree of PV stenosis by peak gradient across the PV in mmhg preoperatively
PV annulus and PV z-score | One week for preoperative assessment.
  Parameters will be measured include median PV annulus diameter in mm , median PV Z-score diameter in mm preoperatively
degree of PV regurge, degree of TR and RV size | One week for preoperative assessment.
  Parameters will be measured include degree of PV regurge jet size by color doppler,degree of TR by jet area -central jets in cm^2 , RV size (RV diastolic area in cm^ , RV systolic area in cm^ ) preoperatively
Age | One week for preoperative assessment
  Parameters will be measured include age in months preoperatively

SECONDARY OUTCOMES:
Gender | Pre-discharge postoperative assessment within one month
  Parameters will be measured include gender pre-discharge postoperative assessment.
Body weight | Pre-discharge postoperative assessment within one month
  Parameters will be measured include body weight in kilograms pre-discharge postoperative assessment.
Height | Pre-discharge postoperative assessment within one month
  Parameters will be measured include height in meters pre-discharge postoperative assessment.
Oxygen saturation , RV function | Pre-discharge postoperative assessment within one month
  Parameters will be measured include Oxygen saturation level % , RV function by measure RV fractional area changes (RVFAC) % Pre-discharge postoperative assessment.
Median RVOT gradient and degree of PV stenosis | Pre-discharge postoperative assessment within one month
  Parameters will be measured include median RVOT gradient in mmhg , degree of PV stenosis by peak gradient across the PV in mmhg pre-discharge postoperative assessment.
PV annulus and PV z-score | Pre-discharge postoperative assessment within one month
  Parameters will be measured include median PV annulus diameter in mm , median PV Z-score diameter in mm pre-discharge postoperative assessment.
degree of PV regurge, degree of TR and RV size | Pre-discharge postoperative assessment within one month
  Parameters will be measured include degree of PV regurge jet size by color doppler,degree of TR by jet area -central jets in cm^2 , RV size (RV diastolic area in cm^ , RV systolic area in cm^ ) pre-discharge postoperative assessment.
Median cross clamp time and CPB time | Pre-discharge postoperative assessment within one month
  Parameters will be measured include Median cross clamp time in minutes and CPB time in minutes pre-discharge postoperative assessment.
ICU stay | Pre-discharge postoperative assessment within one month
  Parameters will be measured include ICU stay days pre-discharge postoperative assessment.
Time till weaning from mechanical ventilator | Pre-discharge postoperative assessment within one month
  Parameters will be measured include Time till weaning from mechanical ventilator in hours pre-discharge postoperative assessment.
Age | Pre-discharge postoperative assessment within one month
  Parameters will be measured include age in months pre-discharge postoperative assessment.

OTHER OUTCOMES:
Gender | Reassessment after 6 months.
  Parameters will be measured include gender in follow up after 6 months.
Body weight | Reassessment after 6 months.
  Parameters will be measured include body weight in kilograms in follow up after 6 months.
Height | Reassessment after 6 months.
  Parameters will be measured include body height in meters in follow up after 6 months.
Oxygen saturation , RV function | Reassessment after 6 months.
  Parameters will be measured include Oxygen saturation level % , RV function by measure RV fractional area changes (RVFAC) % in follow up after 6 months.
include median RVOT gradient and degree of PV stenosis | Reassessment after 6 months.
  Parameters will be measured include include median RVOT gradient in mmhg and degree of PV stenosis by peak gradient across the PV in mmhg in follow up after 6 months.
PV annulus and PV z-score | Reassessment after 6 months.
  Parameters will be measured include median PV annulus diameter in mm , median PV Z-score diameter in mm in follow up after 6 months.
degree of PV regurge, degree of TR and RV size | Reassessment after 6 months.
  Parameters will be measured include degree of PV regurge jet size by color doppler,degree of TR by jet area -central jets in cm^2 , RV size (RV diastolic area in cm^ , RV systolic area in cm^ ) in follow up after 6 months.
Age | Reassessment after 6 months.
  Parameters will be measured include age in months in follow up after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M. El-Minshawy, Prof, Study Chair — Assiut University; Mahmoud Kh Abdelatif, Ass.lecturer, Study Director — Assiut University

REFERENCES:
- [Background] Kwak JG, Kim WH, Kim ER, Lim JH, Min J. One-Year Follow-up After Tetralogy of Fallot Total Repair Preserving Pulmonary Valve and Avoiding Right Ventriculotomy. Circ J. 2018 Nov 24;82(12):3064-3068. doi: 10.1253/circj.CJ-18-0690. Epub 2018 Oct 5. PMID 30298850
- [Background] Vida VL, Angelini A, Guariento A, Frescura C, Fedrigo M, Padalino M, Sanders SP, Thiene G, Stellin G. Preserving the pulmonary valve during early repair of tetralogy of Fallot: Anatomic substrates and surgical strategies. J Thorac Cardiovasc Surg. 2015 May;149(5):1358-63.e1. doi: 10.1016/j.jtcvs.2015.01.030. Epub 2015 Jan 21. PMID 25983249